CLINICAL TRIAL: NCT01175044
Title: Efficacy of a Dilute Betadine Lavage in the Prevention of Postoperative Infection in Revision Total Knee Arthroplasty
Brief Title: Dilute Betadine Lavage in the Prevention of Postoperative Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Central DuPage Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10031106
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Prosthesis-Related Infections; Arthroplasty
Keywords: Revision; Knee; Arthroplasty; Betadine; Lavage; Infection
MeSH Terms: conditions — Prosthesis-Related Infections; Infections | interventions — Povidone-Iodine; Therapeutic Irrigation; Second-Look Surgery; Arthroplasty; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Betadine Lavage (Active Comparator): dilute betadine lavage prior to surgical closure for 3 minutes followed by 2000ml of sterile saline irrigation
  Interventions: Procedure: Betadine Lavage
- Saline Lavage (Placebo Comparator): 2000 ml sterile saline lavage alone
  Interventions: Procedure: Saline Lavage

INTERVENTIONS:
Procedure: Betadine Lavage — Following revision knee surgery, a dilute betadine lavage prior to surgical closure for 3 minutes followed by 2000 ml of sterile saline irrigation
  Other Names: Betadine; Lavage; Infection; Revision; Knee; Arthroplasty
  Arms: Betadine Lavage
Procedure: Saline Lavage — Following revision knee surgery, 2000ml sterile saline lavage prior to closure
  Other Names: Saline; Lavage; Infection; Revision; Knee; Arthroplasty
  Arms: Saline Lavage

SUMMARY:
The purpose of this study is to examine the efficacy of a dilute betadine solution in reducing infectious complications in revision total knee arthroplasty. The investigators will enroll patients who are scheduled to undergo a revision total knee arthroplasty. Patients will be randomized into two groups. The treatment group will receive a dilute betadine lavage prior to surgical closure for 3 minutes followed by 2000ml of sterile saline irrigation and the control group will receive the 2000ml sterile saline lavage alone.

DETAILED DESCRIPTION:
Infections in total knee arthroplasty are still a major source of morbidity and mortality in Orthopaedics. They often necessitate long term antibiotics, reoperation, and can lead to further complications such as sepsis or even death. Infection prevention remains one of the primary goals of an orthopedic surgeon. While most sources report the infection rate for primary total knee arthroplasty to be less than 1%, the reported rate for infection in revision total knee arthroplasties has been reported to be as high as 5.6%. Despite steps taken towards infection prevention such as proper administration of preoperative antibiotics, strict adherence to sterile methods, and meticulous sterile preparation of the surgical site; infection remains higher in the total knee revision arthroplasty patient population when compared to primary total knee arthroplasty. A dilute betadine lavage (0.35% to 1% povidone iodine) prior to surgical closure has been shown in general surgical procedures as well as orthopaedic spine surgeries to reduce the infection rate in their patients, but this has not been examined in total joint arthroplasty.

The study will enroll patients who are scheduled to undergo a revision total knee arthroplasty. Patients will be randomized into two groups. The treatment group will receive a dilute betadine lavage prior to surgical closure for 3 minutes followed by 2000ml of sterile saline irrigation and the control group will receive the 2000ml sterile saline lavage alone. All other treatment will be standard of care.

Subjects will then be followed for one year post surgery for infection, as defined by Appendix 1, at intervals of 2 weeks, 6 weeks, 3 months, and one year from the date of surgery. During these visits patients will receive standard post operative care which includes infection screening. If an infection is clinically suspected with symptoms such as warmth and erythema over the joint, reduced mobility of the joint, and increasing pain at the joint, then infection data will be collected which will consist of a Erythrocyte Sedimentation Rate, C-Reactive Protein levels and a synovial fluid sample will be taken for white blood cell count and bacterial culture.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo revision total knee arthroplasty

Exclusion Criteria:

* Inability to provide informed consent or to comply with study assessments (e.g. due to cognitive impairment or geographic distance).
* Age ≤ 17.
* Allergy to povidone iodine.
* Any condition requiring antibiotics 14 days prior to arriving for surgery.
* Patients with chronic immunosuppression (such as HIV/AIDS).
* Unable to adhere to follow up schedule and treatment.
* Patients scheduled to undergo revision total knee arthroplasty for infectious reasons.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Infection Rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Craig J Della Valle, MD, Principal Investigator — Rush University Medical Center
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Central DuPage Hospital, Winfield, Illinois